CLINICAL TRIAL: NCT03835962
Title: Empirical Distributions of ERP Components Elicited by the NeuroCatch™ Platform: Development of a Reference Interval Database
Brief Title: Development of a Reference Interval Database With the NeuroCatch™ Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCI_NCClin_002
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Brain Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): All participants will be asked to attend one experimental session. During the session, participants will listen one auditory stimulus sequence including sounds and words while EEG activity is recorded using the NeuroCatch Platform™ device.
  Interventions: Device: NeuroCatch™ Platform

INTERVENTIONS:
Device: NeuroCatch™ Platform — NeuroCatch Platform™ consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP) information.

SUMMARY:
The NeuroCatch Platform™, an investigational medical device system developed by NeuroCatch Inc., consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP; brain response to a stimulus) information.

The purpose of the study is to understand how the brain responds to sounds and words, and how this response varies between individuals of different age groups. Interindividual variation reflects the many different factors which cause results to vary from one individual to another within a population. The current clinical study aims to establish a reference interval database of ERPs. These reference intervals will characterize the expected range of interindividual variability between groups. Reference interval databases provide a tool for comparing the results from one individual with those from other members of the same age group.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex, at least 8 years of age or older
2. Able to understand the informed consent/assent form, study procedures and willing to participate in study
3. Able to remain seated and focused for 6 minutes
4. Normal hearing capabilities

Exclusion Criteria:

1. Clinically documented hearing issues (e.g. tinnitus, in-ear hearing problems or punctured ear drum)
2. Implanted pacemaker or implanted electrical stimulators
3. Metal or plastic implants in skull
4. Exposed to an investigational drug or device 30 days prior to start in this study, or concurrent or planned use of investigational drug or device while enrolled in this study
5. Not proficient in English language
6. Previous exposure to the NeuroCatch™ Platform audio sequences in the last 6 months
7. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
8. History of seizures
9. Allergy to rubbing alcohol or EEG gel
10. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin)

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Response size of selected ERPs (N100, P300, N400) acquired using the NeuroCatch™ Platform | 1 day
  Response size will be measured as amplitude in microvolts.
Response timing of selected ERPs (N100, P300, N400) acquired using the NeuroCatch™ Platform | 1 day
  Response timing will be measured as latency in milliseconds.

SECONDARY OUTCOMES:
Collection and evaluation of adverse events and adverse device effects | 1 day
  Evaluation of safety and tolerability of the NeuroCatch™ Platform device
Demographic indicators (date of birth, sex, level of education, recent sleep, average sleep, fatigue level, recent exercise, recent diet, handedness, first language, medical history, neurological status, and profession) | 1 day
  Secondary statistical analyses will explore relationships between demographic indicators, medical history, neurological status and ERP measures across the sample and within groups.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthTech Connex Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided